CLINICAL TRIAL: NCT01850342
Title: Effectiveness and Safety of Cell-Assisted Lipotransfer for the Treatment of Stress Urinary Incontinence Via Endoscopically-Assisted Administration of Fat Tissue Micrografts Enriched by Autologous Adipose-Derived Regenerative Cells
Brief Title: Effectiveness and Safety of Cell-Assisted Lipotransfer for the Treatment of Stress Urinary Incontinence
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Burnasyan Federal Medical Biophysical Center (Other Government)
Responsible Party: Principal Investigator, Pavel Kyzlasov, MD, Burnasyan Federal Medical Biophysical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-FMBC-01-01-13
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Stress Urinary Incontinence
Keywords: Male stress urinary incontinence; Cell-assisted lipotransfer; Adipose-derived regenerative cells; ADRC; Micrograft; Fat tissue; Stem cells
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fat micrograft enhanced with ADRC (Experimental)
  Interventions: Procedure: Periurethral injection of fat micrograft enriched with ADRC

INTERVENTIONS:
Procedure: Periurethral injection of fat micrograft enriched with ADRC — Subjects will undergo liposuction under local anesthesia. One part of lipoaspirate will be processed to isolate and concentrate ADRCs. Another part of lipoaspirate will be washed and homogenized to prepare fat tissue micrograft. After that fat tissue micrograft will be mixed with ADRC. Autologous fat micrograft enriched with ADRC will be injected at the bulbomembranous region of urethra circle-wise under endoscopic vision.

SUMMARY:
Autologous washed and homogenized fat micrograft harvested from the patient's front abdominal wall enriched with adipose-derived regenerative cells (ADRC) derived by enzyme-treatment of a portion of the harvested fat. Fat tissue micrograft mixed with ADRC will be administered one-time endoscopically into submucosal layer of urethra under eye control. This is a single arm study with no control. All patients receive cell therapy.

DETAILED DESCRIPTION:
Fat tissue obtainment. Subjects will undergo liposuction under local anesthesia. In this procedure, Ringer's solution with the anesthetic lidocaine and vasoconstrictor adrenaline infused into the adipose compartment to minimize blood loss and contamination of the tissue by peripheral blood cells. 15 minutes later a hollow blunt-tipped 3 mm cannula introduced into the subcutaneous space through small (0.5 cm) incision. The cannula attached to syringe and under gentle suction moved through the adipose compartment, mechanically disrupting the fat tissue. Aspirate volume - approximately 150 cc. Procedure time - 30 minutes.

ADRC isolation. Aspirated fat tissue placed into sterile tubes with transport medium and delivered into the laboratory within 15 minutes. To isolate the ADRC, part of lipoaspirate (approximately 100 cc) washed extensively with equal volumes of phosphate-buffered saline and digested with collagenase. After enzyme activity neutralization decomposed fat tissue eliminated and ADRC washed 3 times with saline. Cells divided into 3 portions. First portion used for counting, viability and sterility assessment. Second portion prepared for freezing in liquid nitrogen. Third portion mixed with fat micrograft.

Fat tissue enriched micrograft preparation. Obtained fat tissue (approximately 20-30 cc) washed repeatedly. Aspirated fat settled down in syringes placed in vertical position, after that liquid fraction eliminated. Syringes with fat filled up with Ringer's solution and procedure of settlement repeated 3-5 times. Washed fat placed on metallic mesh and mashed up using metallic spatula. Homogenized fat mixed with prepared ADRC and collected in syringe for further injection. Ratio fat micrograft/fat for ADRC estimated according to aspirate volume and usually forms 1:10. For example, ADRC obtained from 100 cc of fat tissue should be mixed with 10 cc of fat micrograft.

Fat micrograft preparation is also possible in Puregraft System (Cytori Therapeutics Inc) - closed disposable system for fat tissue selective washing.

Periurethral injection of fat micrograft enriched with ADRC Urethra punctured several times circle-wise at the bulbomembranous region at a depth of 5 mm under endoscopic vision and 0.5-1 mL of fat micrograft enriched with ADRC injected each time. Total volume of solution injected - approximately 8 mL. After fat micrograft injected, urethral balloon catheter placed and removed the following day.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffers from stress urinary incontinence due to insufficiency of the urethral sphincter at least for 2 years.
* Moderate and severe grade of urinary incontinence according to assessment made by investigator.
* Patient is familiar with Participant information sheet.
* Patient signed informed consent form.

Exclusion Criteria:

* Contraindications for local anesthesia.

For the patients undergone surgical treatment of prostate cancer:

* Cancer relapse.
* prostate-specific antigen (PSA) level >0.008 ng/mL.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-03 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints | 4 weeks after treatment
  Types, probability and severity of treatment emergent serious adverse events (SAEs) and serious adverse reactions (SARs)

SECONDARY OUTCOMES:
Efficacy endpoints | 2, 4, 8, 12, 16, 24 weeks after treatment
  1. 24-hours pad test
  2. Urodynamic studies: maximal urethral closure pressure (MUCP), functional profile length (FPL), postvoid residual (PVR) volume measurement, uroflowmetry.
  3. Quality of life measured by the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF).

CONTACTS AND LOCATIONS:
Overall Officials: Ilya I Eremin, MD, PhD, Principal Investigator — Burnasyan Federal Medical Biophysical Center; Pavel S Kyzlasov, MD, Principal Investigator — Burnasyan Federal Medical Biophysical Center
Locations (1):
- State Research Center Burnasyan Federal Medical Biophysical Center FMBA of Russia; Center for Biomedical Technologies, Moscow, Russia